CLINICAL TRIAL: NCT03835975
Title: A PHASE 3, RANDOMIZED, OPEN-LABEL TRIAL TO EVALUATE THE SAFETY AND IMMUNOGENICITY OF A 20-VALENT PNEUMOCOCCAL CONJUGATE VACCINE IN ADULTS ≥65 YEARS OF AGE WITH PRIOR PNEUMOCOCCAL VACCINATION
Brief Title: Trial to Evaluate the Safety and Immunogenicity of a 20-Valent Pneumococcal Vaccine in Adults 65 Years of Age or Older With Prior Pneumococcal Vaccination
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: B7471006; 2018-004278-91 (EudraCT Number)
Record Dates: First submitted 2019-02-07; First posted 2019-02-11 (Actual); Results first posted 2021-02-21 (Actual); Last update posted 2021-02-21 (Actual); Status verified 2021-02

CONDITIONS: Pneumococcal Disease
MeSH Terms: conditions — Pneumococcal Infections | interventions — 23-valent pneumococcal capsular polysaccharide vaccine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- 13vPnC (Active Comparator): Pneumococcal conjugate vaccine
  Interventions: Biological: 13vPnC
- PPSV23 (Active Comparator): Pneumococcal polysaccharide vaccine
  Interventions: Biological: PPSV23
- 20vPnC (Experimental): Pneumococcal conjugate vaccine
  Interventions: Biological: 20vPnC

INTERVENTIONS:
Biological: 13vPnC — Pneumococcal conjugate vaccine
  Arms: 13vPnC
Biological: PPSV23 — Pneumococcal polysaccharide vaccine
  Arms: PPSV23
Biological: 20vPnC — Pneumococcal conjugate vaccine
  Arms: 20vPnC

SUMMARY:
This Phase 3 will describe the safety and immunogenicity of a 20-valent pneumococcal conjugate vaccine formulation in adults 65 years of age or older with prior pneumococcal vaccination

ELIGIBILITY:
Inclusion Criteria

1. Male or female adults 65 years of age or greater.
2. Adults determined by clinical assessment, including medical history and clinical judgment, to be eligible for the study, including adults with preexisting stable disease, defined as disease not requiring significant change in therapy in the previous 6 weeks or hospitalization for worsening disease within 12 weeks before receipt of investigational product.
3. Female subject of nonchildbearing potential; male subject not able to father children or who is able to father children and willing to use a highly effective method of contraception.
4. Male or female adults who meet 1 of the following:

   1. Vaccination with PPSV23 greater than or equal to 1 year and less than or equal to 5 years prior to vaccination in the study, and no prior 13vPnC vaccination (Cohort A).
   2. Vaccination with 13vPnC greater than or equal to 6 months prior to vaccination in the study, and no prior PPSV23 vaccination (Cohort B).
   3. Vaccination with 13vPnC followed by PPSV23 (PPSV23 vaccination greater than or equal to 1 year prior to vaccination in the study) (Cohort C).

Exclusion Criteria

1. Serious chronic disorder including metastatic malignancy, severe chronic obstructive pulmonary disease (COPD) requiring supplemental oxygen, end-stage renal disease with or without dialysis, clinically unstable cardiac disease, or any other disorder that, in the investigator's opinion, excludes the subject from participating in the study.
2. History of microbiologically proven invasive disease caused by S pneumoniae.

Min Age: 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 875 (Actual)
Dates: Start 2019-02-12 (Actual); Primary Completion 2020-02-12 (Actual); Study Completion 2020-02-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (41):
- United States (33):
  - Coastal Clinical Research, Inc., Mobile, Alabama
  - East Valley Gastroenterology and Hepatology Associates, Chandler, Arizona
  - The Pain Center of Arizona, Peoria, Arizona
  - HOPE Research Institute, Phoenix, Arizona
  - The Pain Center of Arizona, Phoenix, Arizona
  - Anaheim Clinical Trials, LLC, Anaheim, California
  - Diablo Clinical Research, Inc., Walnut Creek, California
  - Clinical Research Consulting, LLC, Milford, Connecticut
  - Optimal Research, LLC, Melbourne, Florida
  - Synexus Clinical Research US, Inc, The Villages, Florida
  - Meridian Clinical Research, LLC, Savannah, Georgia
  - Clinical Research Atlanta, Stockbridge, Georgia
  - East-West Medical Research Institute, Honolulu, Hawaii
  - Heartland Research Associates, LLC, Wichita, Kansas
  - MedPharmics, LLC, Metairie, Louisiana
  - Meridian Clinical Research, LLC, Rockville, Maryland
  - Meridian Clinical Research, LLC, Norfolk, Nebraska
  - MedPharmics, LLC, Albuquerque, New Mexico
  - Carolina Institute for Clinical Research, Fayetteville, North Carolina
  - PMG Research of Wilmington, LLC, Wilmington, North Carolina
  - CTI Clinical Research Center, Cincinnati, Ohio
  - Sterling Research Group, Ltd., Cincinnati, Ohio
  - Prestige Clinical Research, Franklin, Ohio
  - Lynn Health Science Institute, Oklahoma City, Oklahoma
  - Kaiser Permanente Center For Health Research, Portland, Oregon
  - Columbia Research Group, Inc., Portland, Oregon
  - Medical Research South, LLC, Goose Creek, South Carolina
  - Ventavia Research Group, Keller, Texas
  - J. Lewis Research Inc. / Foothill Family Clinic Draper, Draper, Utah
  - J. Lewis Research, Inc. - Foothill Family Clinic, Salt Lake City, Utah
  - J. Lewis Research, Inc. / Foothill Family Clinic South, Salt Lake City, Utah
  - J. Lewis Research, Inc. / Jordan River Family Medicine, South Jordan, Utah
  - Kaiser Permanente Washington Health Research Institute, Seattle, Washington
- Sweden (8):
  - PharmaSite, Malmo, Skåne County
  - Ladulaas Kliniska Studier, Borås
  - Infektionskliniken, Eskilstuna
  - CTC Gothia Forum, Gothenburg
  - ProbarE i Lund, Lund
  - Avdelningen for Kliniska Provningar, Örebro
  - Karolinska Trial Alliance, KTA Prim, Stockholm
  - Akardo Med Site, Stockholm

IPD SHARING:
Plan to Share IPD: Yes
Pfizer will provide access to individual de-identified participant data and related study documents (e.g. protocol, Statistical Analysis Plan (SAP), Clinical Study Report (CSR)) upon request from qualified researchers, and subject to certain criteria, conditions, and exceptions. Further details on Pfizer's data sharing criteria and process for requesting access can be found at: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests.
URL: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests

REFERENCES:
- [Derived] Cannon K, Elder C, Young M, Scott DA, Scully IL, Baugher G, Peng Y, Jansen KU, Gruber WC, Watson W. A trial to evaluate the safety and immunogenicity of a 20-valent pneumococcal conjugate vaccine in populations of adults >/=65 years of age with different prior pneumococcal vaccination. Vaccine. 2021 Dec 17;39(51):7494-7502. doi: 10.1016/j.vaccine.2021.10.032. Epub 2021 Nov 25. PMID 34839993
- See also: To obtain contact information for a study center near you, click here. — https://pmiform.com/clinical-trial-info-request?StudyID=B7471006

RESULTS

PARTICIPANT FLOW:
Groups:
- Cohort A: 20vPnC: Participants with receipt of 23-valent pneumococcal polysaccharide vaccine (PPSV23) greater than or equal to (>=) 1 to less than or equal to (<=) 5 years, and no 13-valent pneumococcal conjugate vaccine (13vPnC), prior to study vaccination, and randomized to receive a single dose of 0.5 milliliter (mL) intramuscular injection of 20-valent pneumococcal conjugate vaccine (20vPnC) on Day 1.
- Cohort A: 13vPnC: Participants with receipt of PPSV23, >=1 to <=5 years, and no 13vPnC, prior to study vaccination, and randomized to receive a single dose of 0.5 mL intramuscular injection of 13vPnC on Day 1.
- Cohort B: 20vPnC: Participants with receipt of 13vPnC, >=6 months, and no PPSV23, prior to study vaccination, and randomized to receive a single dose of 0.5 mL intramuscular injection of 20vPnC on Day 1.
- Cohort B: PPSV23: Participants with receipt of 13vPnC, >=6 months, and no PPSV23, prior to study vaccination, and randomized to receive a single dose of 0.5 mL intramuscular injection of PPSV23 on Day 1.
- Cohort C: 20vPnC: Participants with receipt of 13vPnC followed by PPSV23 (PPSV23 dose >=1 year) prior to study vaccination, received a single dose of 0.5 mL intramuscular injection of 20vPnC on Day 1.
Period: Overall Study
Arm/Group | Cohort A: 20vPnC | Cohort A: 13vPnC | Cohort B: 20vPnC | Cohort B: PPSV23 | Cohort C: 20vPnC
Started | 253 | 122 | 248 | 127 | 125
Vaccinated | 253 | 122 | 246 | 127 | 125
Safety Population | 253 | 122 | 246 | 127 | 125
Evaluable Immunogenicity Population (for 20vPnC Cohorts) | 247 | 0 | 243 | 0 | 121
Completed | 250 | 119 | 245 | 126 | 125
Not Completed | 3 | 3 | 3 | 1 | 0
Not completed — Lost to Follow-up | 1 | 1 | 0 | 0 | 0
Not completed — No longer met eligibility criteria | 0 | 1 | 0 | 0 | 0
Not completed — Protocol Violation | 1 | 1 | 2 | 0 | 0
Not completed — Withdrawal by Subject | 1 | 0 | 1 | 1 | 0

BASELINE CHARACTERISTICS:
Population: All randomized population.
Groups:
- Total: Total of all reporting groups
Arm/Group | Cohort A: 20vPnC | Cohort A: 13vPnC | Cohort B: 20vPnC | Cohort B: PPSV23 | Cohort C: 20vPnC | Total
Number analyzed (Participants) | 253 | 122 | 248 | 127 | 125 | 875
Age, Continuous [Mean (Standard Deviation); unit: years] | 69.6 (3.88) | 70.2 (4.09) | 70.7 (5.70) | 70.6 (5.73) | 70.8 (4.26) | 70.3 (4.84)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 140 | 64 | 140 | 68 | 65 | 477
  Male | 113 | 58 | 108 | 59 | 60 | 398
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 4 | 3 | 6 | 1 | 2 | 16
  Not Hispanic or Latino | 247 | 117 | 233 | 122 | 113 | 832
  Unknown or Not Reported | 2 | 2 | 9 | 4 | 10 | 27
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 0 | 1 | 0 | 0 | 2
  Asian | 1 | 2 | 0 | 2 | 0 | 5
  Native Hawaiian or Other Pacific Islander | 0 | 1 | 1 | 1 | 0 | 3
  Black or African American | 15 | 8 | 14 | 6 | 4 | 47
  White | 236 | 110 | 228 | 118 | 117 | 809
  More than one race | 0 | 0 | 1 | 0 | 3 | 4
  Unknown or Not Reported | 0 | 1 | 3 | 0 | 1 | 5

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With Local Reactions Within 10 Days After Vaccination
Description: Local reactions were recorded using an electronic diary (e-diary). Local reactions included redness, swelling and pain at the injection site. Redness and swelling were measured and recorded in measuring device units. 1 measuring device unit =0.5 centimeter (cm). Redness and swelling were graded as mild (greater than [>] 2.0 to 5.0 cm), moderate (>5.0 to 10.0 cm) and severe (>10.0 cm). Pain at injection site was graded as mild (did not interfere with activity), moderate (interfered with activity), and severe (prevented daily activity).
Time Frame: Within 10 days after vaccination
Population: The safety population included participants who received 1 dose of 20vPnC, PPSV23, or 13vPnC and had safety follow-up after vaccination. Here, "Overall Number of Participants Analyzed" refers to number of participants with any e-diary data reported after vaccination in the safety population.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Cohort A: 20vPnC | Cohort A: 13vPnC | Cohort B: 20vPnC | Cohort B: PPSV23 | Cohort C: 20vPnC
Number analyzed (Participants) | 253 | 121 | 245 | 126 | 125
percentage of participants
  Redness: Any | 7.9 [4.9 to 11.9] | 2.5 [0.5 to 7.1] | 8.6 [5.4 to 12.8] | 12.7 [7.4 to 19.8] | 4.8 [1.8 to 10.2]
  Redness: Mild | 3.6 [1.6 to 6.6] | 1.7 [0.2 to 5.8] | 2.9 [1.2 to 5.8] | 4.8 [1.8 to 10.1] | 1.6 [0.2 to 5.7]
  Redness: Moderate | 3.2 [1.4 to 6.1] | 0.8 [0.0 to 4.5] | 5.3 [2.9 to 8.9] | 7.1 [3.3 to 13.1] | 3.2 [0.9 to 8.0]
  Redness: Severe | 1.2 [0.2 to 3.4] | 0 [0.0 to 3.0] | 0.4 [0.0 to 2.3] | 0.8 [0.0 to 4.3] | 0 [0.0 to 2.9]
  Swelling: Any | 9.9 [6.5 to 14.2] | 6.6 [2.9 to 12.6] | 9.4 [6.0 to 13.8] | 14.3 [8.7 to 21.6] | 4.0 [1.3 to 9.1]
  Swelling: Mild | 5.1 [2.8 to 8.6] | 6.6 [2.9 to 12.6] | 5.7 [3.2 to 9.4] | 6.3 [2.8 to 12.1] | 1.6 [0.2 to 5.7]
  Swelling: Moderate | 3.6 [1.6 to 6.6] | 0 [0.0 to 3.0] | 3.7 [1.7 to 6.9] | 7.1 [3.3 to 13.1] | 2.4 [0.5 to 6.9]
  Swelling: Severe | 1.2 [0.2 to 3.4] | 0 [0.0 to 3.0] | 0 [0.0 to 1.5] | 0.8 [0.0 to 4.3] | 0 [0.0 to 2.9]
  Pain at the injection site: Any | 50.2 [43.9 to 56.5] | 43.0 [34.0 to 52.3] | 61.2 [54.8 to 67.4] | 56.3 [47.2 to 65.2] | 52.8 [43.7 to 61.8]
  Pain at the injection site: Mild | 45.8 [39.6 to 52.2] | 38.8 [30.1 to 48.1] | 54.7 [48.2 to 61.0] | 40.5 [31.8 to 49.6] | 47.2 [38.2 to 56.3]
  Pain at the injection site: Moderate | 4.3 [2.2 to 7.6] | 3.3 [0.9 to 8.2] | 6.1 [3.5 to 9.9] | 14.3 [8.7 to 21.6] | 5.6 [2.3 to 11.2]
  Pain at the injection site: Severe | 0 [0.0 to 1.4] | 0.8 [0.0 to 4.5] | 0.4 [0.0 to 2.3] | 1.6 [0.2 to 5.6] | 0 [0.0 to 2.9]

2. Primary Outcome: Percentage of Participants With Systemic Events Within 7 Days After Vaccination
Description: Systemic events fever, fatigue, headache, muscle pain and joint pain were recorded by using an e-diary. Fever was defined as temperature >=38.0 degree Celsius (C) and categorized to >=38.0 to 38.4 degree C, >38.4 to 38.9 degree C, >38.9 to 40.0 degree C and >40.0 degree C. Fatigue, headache, muscle pain and joint pain were graded as mild (did not interfere with activity), moderate (some interference with activity) and severe (prevented daily routine activity).
Time Frame: Within 7 days after vaccination
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Cohort A: 20vPnC | Cohort A: 13vPnC | Cohort B: 20vPnC | Cohort B: PPSV23 | Cohort C: 20vPnC
Number analyzed (Participants) | 253 | 121 | 245 | 126 | 125
percentage of participants
  Fever: >=38.0 degree C | 0.8 [0.1 to 2.8] | 0 [0.0 to 3.0] | 0 [0.0 to 1.5] | 1.6 [0.2 to 5.6] | 0 [0.0 to 2.9]
  Fever: >=38.0 degree C to 38.4 degree C | 0.8 [0.1 to 2.8] | 0 [0.0 to 3.0] | 0 [0.0 to 1.5] | 0.8 [0.0 to 4.3] | 0 [0.0 to 2.9]
  Fever: >38.4 degree C to 38.9 degree C | 0 [0.0 to 1.4] | 0 [0.0 to 3.0] | 0 [0.0 to 1.5] | 0.8 [0.0 to 4.3] | 0 [0.0 to 2.9]
  Fever: >38.9 degree C to 40.0 degree C | 0 [0.0 to 1.4] | 0 [0.0 to 3.0] | 0 [0.0 to 1.5] | 0 [0.0 to 2.9] | 0 [0.0 to 2.9]
  Fever: >40.0 degree C | 0 [0.0 to 1.4] | 0 [0.0 to 3.0] | 0 [0.0 to 1.5] | 0 [0.0 to 2.9] | 0 [0.0 to 2.9]
  Fatigue: Any | 28.9 [23.4 to 34.9] | 22.3 [15.2 to 30.8] | 31.0 [25.3 to 37.2] | 33.3 [25.2 to 42.3] | 32.8 [24.7 to 41.8]
  Fatigue: Mild | 17.8 [13.3 to 23.1] | 9.9 [5.2 to 16.7] | 19.6 [14.8 to 25.1] | 19.8 [13.3 to 27.9] | 19.2 [12.7 to 27.2]
  Fatigue: Moderate | 11.1 [7.5 to 15.6] | 9.9 [5.2 to 16.7] | 10.2 [6.7 to 14.7] | 13.5 [8.1 to 20.7] | 12.0 [6.9 to 19.0]
  Fatigue: Severe | 0 [0.0 to 1.4] | 2.5 [0.5 to 7.1] | 1.2 [0.3 to 3.5] | 0 [0.0 to 2.9] | 1.6 [0.2 to 5.7]
  Headache: Any | 17.8 [13.3 to 23.1] | 18.2 [11.8 to 26.2] | 13.5 [9.5 to 18.4] | 21.4 [14.6 to 29.6] | 19.2 [12.7 to 27.2]
  Headache: Mild | 12.6 [8.8 to 17.4] | 12.4 [7.1 to 19.6] | 9.8 [6.4 to 14.2] | 20.6 [13.9 to 28.8] | 12.8 [7.5 to 20.0]
  Headache: Moderate | 4.7 [2.5 to 8.1] | 5.8 [2.4 to 11.6] | 3.7 [1.7 to 6.9] | 0.8 [0.0 to 4.3] | 5.6 [2.3 to 11.2]
  Headache: Severe | 0.4 [0.0 to 2.2] | 0 [0.0 to 3.0] | 0 [0.0 to 1.5] | 0 [0.0 to 2.9] | 0.8 [0.0 to 4.4]
  Muscle Pain: Any | 32.0 [26.3 to 38.1] | 31.4 [23.3 to 40.5] | 33.9 [28.0 to 40.2] | 46.0 [37.1 to 55.1] | 37.6 [29.1 to 46.7]
  Muscle Pain: Mild | 26.1 [20.8 to 32.0] | 24.0 [16.7 to 32.6] | 25.3 [20.0 to 31.2] | 31.7 [23.7 to 40.6] | 28.0 [20.3 to 36.7]
  Muscle Pain: Moderate | 5.5 [3.1 to 9.1] | 5.0 [1.8 to 10.5] | 8.6 [5.4 to 12.8] | 11.9 [6.8 to 18.9] | 8.8 [4.5 to 15.2]
  Muscle Pain: Severe | 0.4 [0.0 to 2.2] | 2.5 [0.5 to 7.1] | 0 [0.0 to 1.5] | 2.4 [0.5 to 6.8] | 0.8 [0.0 to 4.4]
  Joint Pain: Any | 6.7 [4.0 to 10.5] | 10.7 [5.8 to 17.7] | 11.8 [8.1 to 16.6] | 15.9 [10.0 to 23.4] | 16.8 [10.7 to 24.5]
  Joint Pain: Mild | 4.7 [2.5 to 8.1] | 5.0 [1.8 to 10.5] | 7.8 [4.7 to 11.8] | 10.3 [5.6 to 17.0] | 12.8 [7.5 to 20.0]
  Joint Pain: Moderate | 2.0 [0.6 to 4.6] | 5.0 [1.8 to 10.5] | 4.1 [2.0 to 7.4] | 5.6 [2.3 to 11.1] | 4.0 [1.3 to 9.1]
  Joint Pain: Severe | 0 [0.0 to 1.4] | 0.8 [0.0 to 4.5] | 0 [0.0 to 1.5] | 0 [0.0 to 2.9] | 0 [0.0 to 2.9]

3. Primary Outcome: Percentage of Participants With Adverse Events (AEs) Within 1 Month After Vaccination
Description: An AE was any untoward medical occurrence in study participants who received study vaccine without regard to possibility of causal relationship with the treatment.
Time Frame: Within 1 month after vaccination
Population: The safety population included participants who received 1 dose of 20vPnC, PPSV23, or 13vPnC and had safety follow-up after vaccination.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Cohort A: 20vPnC | Cohort A: 13vPnC | Cohort B: 20vPnC | Cohort B: PPSV23 | Cohort C: 20vPnC
Number analyzed (Participants) | 253 | 122 | 246 | 127 | 125
percentage of participants | 7.5 [4.6 to 11.5] | 9.0 [4.6 to 15.6] | 4.9 [2.5 to 8.4] | 11.0 [6.2 to 17.8] | 10.4 [5.7 to 17.1]

4. Primary Outcome: Percentage of Participants With Serious Adverse Events (SAEs) Within 6 Months After Vaccination
Description: An SAE was any untoward medical occurrence at any dose that results in death; is life-threatening (immediate risk of death); requires inpatient hospitalization or prolongation of existing hospitalization; results in persistent or significant disability/incapacity (substantial disruption of the ability to conduct normal life functions); results in congenital anomaly/birth defect or that is considered to be an important medical event.
Time Frame: Within 6 months after vaccination
Population: as for outcome 3
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Cohort A: 20vPnC | Cohort A: 13vPnC | Cohort B: 20vPnC | Cohort B: PPSV23 | Cohort C: 20vPnC
Number analyzed (Participants) | 253 | 122 | 246 | 127 | 125
percentage of participants | 0.8 [0.1 to 2.8] | 1.6 [0.2 to 5.8] | 2.4 [0.9 to 5.2] | 1.6 [0.2 to 5.6] | 1.6 [0.2 to 5.7]

5. Primary Outcome: Percentage of Participants With Newly Diagnosed Chronic Medical Conditions (NDCMCs) Within 6 Months After Vaccination
Description: An NDCMC was defined as a disease or medical condition, not previously identified, that was expected to be persistent or was otherwise long-lasting in its effects.
Time Frame: Within 6 months after vaccination
Population: as for outcome 3
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Cohort A: 20vPnC | Cohort A: 13vPnC | Cohort B: 20vPnC | Cohort B: PPSV23 | Cohort C: 20vPnC
Number analyzed (Participants) | 253 | 122 | 246 | 127 | 125
percentage of participants | 2.0 [0.6 to 4.6] | 0.8 [0.0 to 4.5] | 2.8 [1.2 to 5.8] | 2.4 [0.5 to 6.7] | 4.0 [1.3 to 9.1]

6. Primary Outcome: Pneumococcal Opsonophagocytic Activity (OPA) Geometric Mean Titers (GMTs) at 1 Month After Vaccination
Description: OPA GMTs were determined for serotypes: 1, 3, 4, 5, 6A, 6B, 7F, 9V, 14, 18C, 19A, 19F, 23F, 8, 10A, 11A, 12F, 15B, 22F and 33F. OPA titer was expressed as reciprocal of the highest serum dilution.
Time Frame: 1 month after vaccination
Population: Evaluable immunogenicity population: All participants who received 20vPnC as randomized, enrolled in appropriate cohort based on prior vaccination history, had Visit 2 blood collection within 27 to 49 days after vaccination, had at least 1 valid and determinate OPA titer for any serotype for Visit 2, had no major protocol deviations. Data for this outcome measure were planned to be analyzed for 20vPnC groups of each cohort. Number Analyzed =number of participants evaluable for each serotypes.
Measure: Geometric Mean (95% Confidence Interval); unit: titer
Arm/Group | Cohort A: 20vPnC | Cohort B: 20vPnC | Cohort C: 20vPnC
Number analyzed (Participants) | 247 | 243 | 121
titer
  Serotype 1: number analyzed (Participants) | 246 | 243 | 120
  Serotype 1 | 50.8 [41.6 to 62.0] | 115.3 [96.3 to 137.9] | 82.1 [61.2 to 110.1]
  Serotype 3: number analyzed (Participants) | 243 | 242 | 119
  Serotype 3 | 31.1 [26.7 to 36.1] | 54.3 [46.9 to 62.8] | 39.3 [32.0 to 48.2]
  Serotype 4: number analyzed (Participants) | 236 | 241 | 116
  Serotype 4 | 149.9 [118.2 to 190.1] | 334.9 [273.8 to 409.5] | 193.7 [143.2 to 262.0]
  Serotype 5: number analyzed (Participants) | 244 | 243 | 120
  Serotype 5 | 62.8 [52.7 to 74.9] | 87.3 [73.2 to 104.2] | 83.5 [64.8 to 107.6]
  Serotype 6A: number analyzed (Participants) | 242 | 241 | 121
  Serotype 6A | 748.7 [576.7 to 972.0] | 1080.9 [880.2 to 1327.4] | 1085.3 [796.9 to 1478.1]
  Serotype 6B: number analyzed (Participants) | 243 | 241 | 121
  Serotype 6B | 727.3 [573.6 to 922.1] | 1159.4 [950.7 to 1413.8] | 1033.3 [754.6 to 1414.8]
  Serotype 7F: number analyzed (Participants) | 240 | 243 | 120
  Serotype 7F | 378.1 [316.4 to 451.9] | 555.4 [466.8 to 660.9] | 345.8 [277.0 to 431.7]
  Serotype 9V: number analyzed (Participants) | 241 | 237 | 117
  Serotype 9V | 550.3 [454.0 to 666.9] | 1085.0 [893.5 to 1317.5] | 723.4 [558.1 to 937.6]
  Serotype 14: number analyzed (Participants) | 240 | 242 | 119
  Serotype 14 | 391.2 [314.6 to 486.3] | 664.9 [554.1 to 797.9] | 580.5 [433.7 to 777.0]
  Serotype 18C: number analyzed (Participants) | 245 | 240 | 120
  Serotype 18C | 551.9 [445.1 to 684.4] | 845.9 [692.5 to 1033.1] | 621.2 [469.9 to 821.3]
  Serotype 19A: number analyzed (Participants) | 242 | 242 | 120
  Serotype 19A | 238.6 [197.5 to 288.4] | 365.1 [303.0 to 440.0] | 340.6 [264.1 to 439.2]
  Serotype 19F: number analyzed (Participants) | 244 | 242 | 118
  Serotype 19F | 159.0 [131.4 to 192.3] | 242.3 [199.4 to 294.3] | 217.7 [168.1 to 281.8]
  Serotype 23F: number analyzed (Participants) | 245 | 243 | 120
  Serotype 23F | 151.6 [115.3 to 199.3] | 450.2 [357.8 to 566.4] | 292.6 [203.6 to 420.5]
  Serotype 8: number analyzed (Participants) | 230 | 226 | 109
  Serotype 8 | 211.9 [172.0 to 261.0] | 602.9 [482.9 to 752.8] | 293.8 [220.0 to 392.4]
  Serotype 10A: number analyzed (Participants) | 219 | 210 | 110
  Serotype 10A | 1012.1 [806.7 to 1269.8] | 2005.4 [1586.0 to 2535.7] | 1580.3 [1175.9 to 2123.8]
  Serotype 11A: number analyzed (Participants) | 216 | 206 | 102
  Serotype 11A | 1473.2 [1192.4 to 1820.2] | 1908.2 [1541.5 to 2362.2] | 1566.6 [1140.7 to 2151.4]
  Serotype 12F: number analyzed (Participants) | 224 | 214 | 110
  Serotype 12F | 1054.5 [822.0 to 1352.7] | 1763.4 [1371.8 to 2266.7] | 1401.2 [1001.8 to 1959.7]
  Serotype 15B: number analyzed (Participants) | 225 | 201 | 110
  Serotype 15B | 647.1 [490.8 to 853.1] | 1479.5 [1093.0 to 2002.8] | 1066.9 [721.3 to 1578.1]
  Serotype 22F: number analyzed (Participants) | 218 | 206 | 108
  Serotype 22F | 1772.8 [1354.7 to 2319.8] | 4156.5 [3243.8 to 5326.2] | 2717.8 [1978.4 to 3733.4]
  Serotype 33F: number analyzed (Participants) | 216 | 208 | 103
  Serotype 33F | 2026.2 [1684.3 to 2437.4] | 3174.9 [2579.1 to 3908.3] | 2182.9 [1638.6 to 2907.8]

7. Secondary Outcome: Pneumococcal OPA Geometric Mean Fold Rise (GMFR) From Before Vaccination to 1 Month After Vaccination
Description: OPA GMFR is the ratio of OPA GMTs, 1 month after vaccination to before vaccination. OPA GMFRs from before to 1 month after vaccination were calculated for pneumococcal serotypes 1, 3, 4, 5, 6A, 6B, 7F, 9V, 14, 18C, 19A, 19F, 23F, 8, 10A, 11A, 12F, 15B, 22F and 33F.
Time Frame: From before vaccination to 1 month after vaccination
Population: Evaluable immunogenicity population was analyzed. Data for this outcome measure were planned to be analyzed for 20vPnC groups of each cohort. Number analyzed= number of participants evaluable with OPA titers available at both time points for each serotype.
Measure: Geometric Mean (95% Confidence Interval); unit: fold rise
Arm/Group | Cohort A: 20vPnC | Cohort B: 20vPnC | Cohort C: 20vPnC
Number analyzed (Participants) | 247 | 243 | 121
fold rise
  Serotype 1: number analyzed (Participants) | 245 | 243 | 120
  Serotype 1 | 2.2 [1.9 to 2.5] | 3.4 [2.9 to 4.1] | 2.0 [1.7 to 2.4]
  Serotype 3: number analyzed (Participants) | 243 | 240 | 119
  Serotype 3 | 2.4 [2.1 to 2.8] | 3.5 [3.1 to 4.1] | 1.9 [1.6 to 2.3]
  Serotype 4: number analyzed (Participants) | 231 | 235 | 115
  Serotype 4 | 4.9 [3.9 to 6.1] | 5.0 [4.1 to 6.2] | 2.4 [1.9 to 3.1]
  Serotype 5: number analyzed (Participants) | 241 | 243 | 120
  Serotype 5 | 2.3 [2.0 to 2.6] | 2.3 [2.0 to 2.6] | 1.8 [1.5 to 2.0]
  Serotype 6A: number analyzed (Participants) | 239 | 234 | 118
  Serotype 6A | 12.6 [9.5 to 16.7] | 8.3 [6.6 to 10.4] | 6.5 [4.7 to 9.1]
  Serotype 6B: number analyzed (Participants) | 238 | 238 | 119
  Serotype 6B | 6.6 [5.2 to 8.4] | 6.7 [5.4 to 8.3] | 4.0 [3.0 to 5.2]
  Serotype 7F: number analyzed (Participants) | 233 | 241 | 119
  Serotype 7F | 2.3 [1.9 to 2.7] | 2.6 [2.2 to 3.0] | 1.6 [1.4 to 2.0]
  Serotype 9V: number analyzed (Participants) | 226 | 228 | 114
  Serotype 9V | 2.4 [2.1 to 2.9] | 3.1 [2.6 to 3.6] | 2.1 [1.7 to 2.6]
  Serotype 14: number analyzed (Participants) | 236 | 237 | 119
  Serotype 14 | 1.8 [1.5 to 2.1] | 2.3 [1.9 to 2.8] | 1.7 [1.4 to 2.1]
  Serotype 18C: number analyzed (Participants) | 245 | 240 | 119
  Serotype 18C | 3.2 [2.5 to 3.9] | 3.9 [3.2 to 4.8] | 2.2 [1.8 to 2.7]
  Serotype 19A: number analyzed (Participants) | 239 | 239 | 117
  Serotype 19A | 2.9 [2.4 to 3.4] | 2.9 [2.4 to 3.4] | 1.9 [1.6 to 2.2]
  Serotype 19F: number analyzed (Participants) | 243 | 241 | 118
  Serotype 19F | 2.6 [2.2 to 3.1] | 2.7 [2.3 to 3.2] | 1.9 [1.5 to 2.3]
  Serotype 23F: number analyzed (Participants) | 242 | 242 | 119
  Serotype 23F | 6.6 [5.1 to 8.5] | 9.3 [7.4 to 11.8] | 4.5 [3.4 to 6.0]
  Serotype 8: number analyzed (Participants) | 223 | 219 | 101
  Serotype 8 | 3.6 [2.9 to 4.4] | 22.5 [17.2 to 29.4] | 2.1 [1.6 to 2.8]
  Serotype 10A: number analyzed (Participants) | 198 | 199 | 109
  Serotype 10A | 4.5 [3.5 to 5.7] | 14.4 [10.9 to 19.0] | 4.4 [3.3 to 6.0]
  Serotype 11A: number analyzed (Participants) | 184 | 183 | 91
  Serotype 11A | 2.5 [2.0 to 3.2] | 6.7 [5.0 to 9.0] | 3.1 [2.2 to 4.4]
  Serotype 12F: number analyzed (Participants) | 208 | 200 | 103
  Serotype 12F | 7.2 [5.5 to 9.5] | 31.7 [23.1 to 43.4] | 3.8 [2.7 to 5.5]
  Serotype 15B: number analyzed (Participants) | 211 | 184 | 99
  Serotype 15B | 4.3 [3.3 to 5.7] | 18.9 [13.0 to 27.4] | 4.8 [3.1 to 7.5]
  Serotype 22F: number analyzed (Participants) | 207 | 191 | 104
  Serotype 22F | 11.1 [8.0 to 15.3] | 66.9 [46.5 to 96.4] | 9.8 [6.2 to 15.6]
  Serotype 33F: number analyzed (Participants) | 203 | 196 | 99
  Serotype 33F | 1.8 [1.5 to 2.2] | 5.4 [4.2 to 6.8] | 1.8 [1.4 to 2.2]

8. Secondary Outcome: Percentage of Participants With >=4-Fold Rise in Pneumococcal OPA Titers From Before Vaccination to 1 Month After Vaccination
Description: Percentage of participants with a >=4-fold rise in pneumococcal OPA titers from before vaccination to 1 month after vaccination were calculated for pneumococcal serotypes 1, 3, 4, 5, 6A, 6B, 7F, 9V, 14, 18C, 19A, 19F, 23F, 8, 10A, 11A, 12F, 15B, 22F and 33F.
Time Frame: From before vaccination to 1 month after vaccination
Population: Evaluable immunogenicity population: All participants who received 20vPnC as randomized, enrolled in appropriate cohort based on prior vaccination history, had Visit 2 blood collection within 27 to 49 days after vaccination, had at least 1 valid and determinate OPA titer for any serotype for Visit 2, had no major protocol deviations. Data for this outcome measure were planned to be analyzed for 20vPnC groups of each cohort. Number Analyzed =number of participants evaluable for each serotype.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Cohort A: 20vPnC | Cohort B: 20vPnC | Cohort C: 20vPnC
Number analyzed (Participants) | 247 | 243 | 121
percentage of participants
  Serotype 1: number analyzed (Participants) | 245 | 243 | 120
  Serotype 1 | 22.9 [17.8 to 28.6] | 40.3 [34.1 to 46.8] | 20.8 [14.0 to 29.2]
  Serotype 3: number analyzed (Participants) | 243 | 240 | 119
  Serotype 3 | 29.6 [24.0 to 35.8] | 41.3 [35.0 to 47.8] | 18.5 [12.0 to 26.6]
  Serotype 4: number analyzed (Participants) | 231 | 235 | 115
  Serotype 4 | 41.1 [34.7 to 47.8] | 41.3 [34.9 to 47.9] | 25.2 [17.6 to 34.2]
  Serotype 5: number analyzed (Participants) | 241 | 243 | 120
  Serotype 5 | 25.7 [20.3 to 31.7] | 27.2 [21.7 to 33.2] | 15.8 [9.8 to 23.6]
  Serotype 6A: number analyzed (Participants) | 239 | 234 | 118
  Serotype 6A | 61.5 [55.0 to 67.7] | 56.4 [49.8 to 62.9] | 44.9 [35.7 to 54.3]
  Serotype 6B: number analyzed (Participants) | 238 | 238 | 119
  Serotype 6B | 53.4 [46.8 to 59.8] | 55.0 [48.5 to 61.5] | 35.3 [26.8 to 44.6]
  Serotype 7F: number analyzed (Participants) | 233 | 241 | 119
  Serotype 7F | 26.2 [20.7 to 32.3] | 30.3 [24.6 to 36.5] | 14.3 [8.5 to 21.9]
  Serotype 9V: number analyzed (Participants) | 226 | 228 | 114
  Serotype 9V | 28.3 [22.5 to 34.7] | 36.0 [29.7 to 42.6] | 20.2 [13.2 to 28.7]
  Serotype 14: number analyzed (Participants) | 236 | 237 | 119
  Serotype 14 | 15.7 [11.3 to 21.0] | 24.9 [19.5 to 30.9] | 16.0 [9.9 to 23.8]
  Serotype 18C: number analyzed (Participants) | 245 | 240 | 119
  Serotype 18C | 29.4 [23.8 to 35.5] | 38.3 [32.2 to 44.8] | 17.6 [11.3 to 25.7]
  Serotype 19A: number analyzed (Participants) | 239 | 239 | 117
  Serotype 19A | 29.7 [24.0 to 35.9] | 29.3 [23.6 to 35.5] | 15.4 [9.4 to 23.2]
  Serotype 19F: number analyzed (Participants) | 243 | 241 | 118
  Serotype 19F | 29.2 [23.6 to 35.4] | 32.8 [26.9 to 39.1] | 16.9 [10.7 to 25.0]
  Serotype 23F: number analyzed (Participants) | 242 | 242 | 119
  Serotype 23F | 49.6 [43.1 to 56.1] | 58.7 [52.2 to 64.9] | 42.9 [33.8 to 52.3]
  Serotype 8: number analyzed (Participants) | 223 | 219 | 101
  Serotype 8 | 39.9 [33.4 to 46.7] | 72.6 [66.2 to 78.4] | 30.7 [21.9 to 40.7]
  Serotype 10A: number analyzed (Participants) | 198 | 199 | 109
  Serotype 10A | 45.5 [38.4 to 52.7] | 70.9 [64.0 to 77.1] | 44.0 [34.5 to 53.9]
  Serotype 11A: number analyzed (Participants) | 184 | 183 | 91
  Serotype 11A | 30.4 [23.9 to 37.6] | 54.6 [47.1 to 62.0] | 35.2 [25.4 to 45.9]
  Serotype 12F: number analyzed (Participants) | 208 | 200 | 103
  Serotype 12F | 51.4 [44.4 to 58.4] | 76.5 [70.0 to 82.2] | 40.8 [31.2 to 50.9]
  Serotype 15B: number analyzed (Participants) | 211 | 184 | 99
  Serotype 15B | 37.4 [30.9 to 44.3] | 66.3 [59.0 to 73.1] | 38.4 [28.8 to 48.7]
  Serotype 22F: number analyzed (Participants) | 207 | 191 | 104
  Serotype 22F | 57.0 [50.0 to 63.8] | 83.2 [77.2 to 88.2] | 54.8 [44.7 to 64.6]
  Serotype 33F: number analyzed (Participants) | 203 | 196 | 99
  Serotype 33F | 18.7 [13.6 to 24.8] | 53.6 [46.3 to 60.7] | 19.2 [12.0 to 28.3]

9. Secondary Outcome: Percentage of Participants With Pneumococcal OPA Titers >=Lower Limit of Quantitation (LLOQ) at 1 Month After Vaccination
Description: The percentage of participants with OPA titers >=LLOQ at 1 month after vaccination were calculated for pneumococcal serotypes 1, 3, 4, 5, 6A, 6B, 7F, 9V, 14, 18C, 19A, 19F, 23F, 8, 10A, 11A, 12F, 15B, 22F and 33F.
Time Frame: 1 month after vaccination
Population: as for outcome 8
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Cohort A: 20vPnC | Cohort B: 20vPnC | Cohort C: 20vPnC
Number analyzed (Participants) | 247 | 243 | 121
percentage of participants
  Serotype 1: number analyzed (Participants) | 246 | 243 | 120
  Serotype 1 | 65.4 [59.1 to 71.4] | 87.7 [82.8 to 91.5] | 77.5 [69.0 to 84.6]
  Serotype 3: number analyzed (Participants) | 243 | 242 | 119
  Serotype 3 | 76.1 [70.3 to 81.3] | 90.5 [86.1 to 93.9] | 87.4 [80.1 to 92.8]
  Serotype 4: number analyzed (Participants) | 236 | 241 | 116
  Serotype 4 | 76.7 [70.8 to 81.9] | 91.7 [87.5 to 94.9] | 87.1 [79.6 to 92.6]
  Serotype 5: number analyzed (Participants) | 244 | 243 | 120
  Serotype 5 | 64.8 [58.4 to 70.7] | 74.9 [69.0 to 80.2] | 72.5 [63.6 to 80.3]
  Serotype 6A: number analyzed (Participants) | 242 | 241 | 121
  Serotype 6A | 84.3 [79.1 to 88.6] | 93.8 [89.9 to 96.5] | 90.9 [84.3 to 95.4]
  Serotype 6B: number analyzed (Participants) | 243 | 241 | 121
  Serotype 6B | 86.8 [81.9 to 90.8] | 93.8 [89.9 to 96.5] | 91.7 [85.3 to 96.0]
  Serotype 7F: number analyzed (Participants) | 240 | 243 | 120
  Serotype 7F | 74.2 [68.1 to 79.6] | 84.8 [79.6 to 89.0] | 79.2 [70.8 to 86.0]
  Serotype 9V: number analyzed (Participants) | 241 | 237 | 117
  Serotype 9V | 76.8 [70.9 to 81.9] | 89.5 [84.8 to 93.1] | 85.5 [77.8 to 91.3]
  Serotype 14: number analyzed (Participants) | 240 | 242 | 119
  Serotype 14 | 85.8 [80.8 to 90.0] | 95.0 [91.5 to 97.4] | 93.3 [87.2 to 97.1]
  Serotype 18C: number analyzed (Participants) | 245 | 240 | 120
  Serotype 18C | 91.8 [87.7 to 94.9] | 96.3 [93.0 to 98.3] | 95.8 [90.5 to 98.6]
  Serotype 19A: number analyzed (Participants) | 242 | 242 | 120
  Serotype 19A | 93.8 [90.0 to 96.5] | 95.9 [92.5 to 98.0] | 98.3 [94.1 to 99.8]
  Serotype 19F: number analyzed (Participants) | 244 | 242 | 118
  Serotype 19F | 71.7 [65.6 to 77.3] | 84.3 [79.1 to 88.6] | 84.7 [77.0 to 90.7]
  Serotype 23F: number analyzed (Participants) | 245 | 243 | 120
  Serotype 23F | 76.3 [70.5 to 81.5] | 93.8 [90.0 to 96.5] | 87.5 [80.2 to 92.8]
  Serotype 8: number analyzed (Participants) | 230 | 226 | 109
  Serotype 8 | 85.2 [80.0 to 89.5] | 94.7 [90.9 to 97.2] | 90.8 [83.8 to 95.5]
  Serotype 10A: number analyzed (Participants) | 219 | 210 | 110
  Serotype 10A | 92.2 [87.9 to 95.4] | 95.7 [92.0 to 98.0] | 96.4 [91.0 to 99.0]
  Serotype 11A: number analyzed (Participants) | 216 | 206 | 102
  Serotype 11A | 91.2 [86.6 to 94.6] | 94.7 [90.6 to 97.3] | 89.2 [81.5 to 94.5]
  Serotype 12F: number analyzed (Participants) | 224 | 214 | 110
  Serotype 12F | 87.9 [82.9 to 91.9] | 93.0 [88.7 to 96.0] | 91.8 [85.0 to 96.2]
  Serotype 15B: number analyzed (Participants) | 225 | 201 | 110
  Serotype 15B | 84.9 [79.5 to 89.3] | 91.0 [86.2 to 94.6] | 90.0 [82.8 to 94.9]
  Serotype 22F: number analyzed (Participants) | 218 | 206 | 108
  Serotype 22F | 94.0 [90.0 to 96.8] | 99.0 [96.5 to 99.9] | 98.1 [93.5 to 99.8]
  Serotype 33F: number analyzed (Participants) | 216 | 208 | 103
  Serotype 33F | 88.9 [83.9 to 92.7] | 91.8 [87.2 to 95.2] | 87.4 [79.4 to 93.1]

ADVERSE EVENTS:
Time Frame: Other AEs: local reactions within 10 days after vaccination, systemic events: within 7 days after vaccination (systematic assessment), non serious AEs up to 1 month after Vaccination; SAEs: up to 6 months after vaccination
Description: Same event may appear as AE and SAE, what is presented are distinct events. Event may be categorized as serious in 1 participant and as non-serious in another participant or 1 participant may have experienced both serious and non-serious event during study. Safety population was analyzed.
Arm/Group | Cohort A: 20vPnC | Cohort A: 13vPnC | Cohort B: 20vPnC | Cohort B: PPSV23 | Cohort C: 20vPnC
All-Cause Mortality (participants affected / at risk) | 0/253 | 0/122 | 0/246 | 0/127 | 0/125
Serious Adverse Events (participants affected / at risk) | 2/253 | 2/122 | 6/246 | 2/127 | 2/125
Other Adverse Events (participants affected / at risk) | 173/253 | 69/122 | 178/246 | 96/127 | 86/125
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Cohort A: 20vPnC (N=253) | Cohort A: 13vPnC (N=122) | Cohort B: 20vPnC (N=246) | Cohort B: PPSV23 (N=127) | Cohort C: 20vPnC (N=125)
Acute myocardial infarction (Cardiac disorders) | 0 | 0 | 1 | 0 | 0
Cardiac failure congestive (Cardiac disorders) | 1 | 0 | 0 | 0 | 0
Dysphagia (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0
Cholecystitis (Hepatobiliary disorders) | 0 | 1 | 0 | 0 | 0
Appendicitis (Infections and infestations) | 0 | 0 | 0 | 1 | 0
Clostridium difficile colitis (Infections and infestations) | 0 | 0 | 0 | 1 | 0
Pneumonia (Infections and infestations) | 0 | 0 | 0 | 0 | 1
Blood pressure decreased (Investigations) | 0 | 1 | 0 | 0 | 0
Dehydration (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1 | 0
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 1
Prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0 | 0
Carotid artery stenosis (Nervous system disorders) | 1 | 0 | 0 | 0 | 0
Syncope (Nervous system disorders) | 0 | 0 | 2 | 0 | 0
Cardiac pacemaker replacement (Surgical and medical procedures) | 0 | 0 | 1 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Cohort A: 20vPnC (N=253) | Cohort A: 13vPnC (N=122) | Cohort B: 20vPnC (N=246) | Cohort B: PPSV23 (N=127) | Cohort C: 20vPnC (N=125)
Fatigue (FATIGUE) (General disorders) | 73 | 27 | 76 | 42 | 41
Injection site erythema (REDNESS) (General disorders) | 20 | 3 | 21 | 16 | 6
Injection site pain (PAIN) (General disorders) | 127 | 52 | 150 | 71 | 66
Injection site swelling (SWELLING) (General disorders) | 25 | 8 | 23 | 18 | 5
Nasopharyngitis (Infections and infestations) | 3 | 1 | 0 | 0 | 0
Urinary tract infection (Infections and infestations) | 0 | 2 | 0 | 0 | 0
Arthralgia (JOINT PAIN) (Musculoskeletal and connective tissue disorders) | 17 | 13 | 29 | 20 | 21
Myalgia (MUSCLE PAIN) (Musculoskeletal and connective tissue disorders) | 81 | 38 | 83 | 58 | 47
Pyrexia (FEVER) (General disorders) | 0 | 0 | 0 | 2 | 0
Dizziness (Nervous system disorders) | 0 | 0 | 1 | 2 | 0
Headache (HEADACHE) (Nervous system disorders) | 45 | 22 | 33 | 27 | 24

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Pfizer has the right to review disclosures, requesting a delay of less than 60 days. Investigator will postpone single center publications until after disclosure of pooled data (all sites), less than 12 months from study completion/termination at all participating sites. Investigator may not disclose previously undisclosed confidential information other than study results.

DOCUMENTS (2):
  • Statistical Analysis Plan (2020-03-23): https://cdn.clinicaltrials.gov/large-docs/75/NCT03835975/SAP_000.pdf
  • Study Protocol (2019-02-11): https://cdn.clinicaltrials.gov/large-docs/75/NCT03835975/Prot_001.pdf